CLINICAL TRIAL: NCT03277716
Title: Effectivity and Safety of Microwave Ablation Combined With Transcatheter Arterial Chemoembolization(TACE) for Huge Unresectable Hepatocellular Carcinoma: a Multicenter Analysis
Brief Title: Microwave Ablation Combined With TACE in the Treatment of Unresectable Huge Hepatocellular Carcinoma Huge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fan Weijun (Other)
Responsible Party: Sponsor-Investigator, Fan Weijun, the professor of Sun Yat-sen University, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sysucc01
Record Dates: First submitted 2017-08-06; First posted 2017-09-11 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Hepatocellular Carcinoma Non-resectable; Transarterial Chemoembolization; Microwave Ablation
Keywords: Huge hepatocellular carcinoma; Microwave ablation; TACE; Safety; Non-resectable; Treatment
MeSH Terms: interventions — Chemoembolization, Therapeutic

STUDY DESIGN:
Intervention Model Description: Microwave Ablation Combined With TACE in the Treatment of Non-resectable Huge Hepatocellular Carcinoma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE+MWA (Experimental): Transcatheter arterial chemoembolization combined with microwave ablation: 2-3 times of TACE treatment, then followed by ablation treatment using MWA system.
  Interventions: Procedure: TACE; Procedure: MWA; Device: MWA system; Drug: Chemoembolization

INTERVENTIONS:
Procedure: TACE — TACE: With the patient under local anesthesia, a 5F French catheter was introduced into the abdominal aorta via the femoral artery using the Seldinger technique. Hepatic arterial angiography was performed using fluoroscopy to guide the catheter into the celiac and superior mesenteric arteries. Then, the feeding arteries, tumor, and vascular anatomy surrounding the tumor were identified. Subsequently, a microcatheter was super-selectively inserted into the feeding arteries. Then, a mixture solution containing chemotherapeutic agents and embolic agents were infused into the artery according to the size and blood supply of the tumors.
  Other Names: Transcatheter arterial chemoembolization procedure
Procedure: MWA — MWA: All patients were instructed to fast from all foods for 12 hours preoperatively. During the procedure, a CT scan was used to locate the liver tumors, and to design the optimal puncture needle route. Routine disinfection and local anesthesia was applied around the puncture point, and a 16-gauge microwave antenna was gradually inserted into the tumor along the pre-determined angle. Settings of the MWA parameters depended on the manufacturer's recommendation and our experience.
  Other Names: Microwave ablation
Device: MWA system — MWA system is a kind of medical treatment instrument to restrain and kill tumor based on microwave heating technique and biology heating effect theory.
  Other Names: Microwave ablation system
Drug: Chemoembolization — Chemotherapeutic drugs: adriamycin，epirubicin and pirarubicin. Embolic agent: lipiodol and embolic microspherea The mixture solution containing chemotherapeutic drugs and embolic agent were infused into the artery according to by the number and size of the lesions, liver and kidney function of the patient, and blood supply of the tumors.
  Other Names: Chemotherapeutic drugs and Embolic agent

SUMMARY:
The purpose of this study was to prospectively evaluate the efficacy and safety of TACE combined with MWA in patients with huge unresectable hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common cancer worldwide. Despite the widespread application of surveillance programs in high-risk populations, patients continue to present with huge (≥ 10 cm) HCCs.And it's still a challenge to treat huge HCC nowadays.Surgical resection is currently the only curative treatment for huge HCCs ; however, only a minority of patients are candidates for curative resection. Sorafenib is recommended for the treatment of advanced HCCs, including huge HCCs, but the usage is severely limited by high adverse event rates and low efficiency. Thus, transarterial chemoembolization (TACE) is considered the first choice for huge unresectable HCCs. Several studies have concluded that TACE effectively improves the overall survival of patients with huge HCCs. Meanwhile, microwave ablation (MWA) now has been shown to be safe and effective for local tumor control in HCC patients. However, neither MWA nor TACE alone can achieve complete control of large HCCs . Therefore, the combination of TACE and MWA (TACE+MWA) is an appealing approach to treat HCCs. TACE+MWA now has been shown to improve overall survival rates compared with TACE alone in patients with small to large HCCs. But little data is available on TACE+MWA in patients with huge unresectable HCCs. Thus, the study was designed.

ELIGIBILITY:
Inclusion Criteria:

1. The performance status of Eastern Cooperative Oncology Group (ECOG) must be 0-1
2. The diagnosis of primary hepatocellular carcinoma must be in line with the American Society for the study of liver diseases (AASLD) diagnostic criteria for hepatocellular carcinoma (HCC)
3. Child-Pugh score A or B;
4. Aged from 18 to 75 years;
5. Subjects voluntarily join the study, and signe informed consent;
6. No anti-tumor therapy was received；
7. Meet the following 4 characteristics: A. primary tumor diameter more than or equal to 10cm; B. no more than 3 HCC foci, and the maximum diameter is less than or equal to 5cm; C. with IIa, I or no portal vein tumor thrombus (Cheng's Classification)；D. the tumor could not be surgically removed
8. No extrahepatic metastases

Exclusion Criteria:

1. Abnormal coagulation function: PLT < 40×109/L, PTA < 40%;
2. Patients have the past history of liver cancer treatment, such as transplantation, resection, radiotherapy, chemotherapy and so on;
3. Patients participated in clinical trials of equipment or drugs (signed informed consent) within 4 weeks;
4. Patients accompany by ascites, hepatic encephalopathy and esophageal and gastric varices bleeding;
5. Any serious accompanying disease, which is expected to have an unknown, impact on the prognosis, include heart disease, inadequately controlled diabetes and psychiatric disorders;
6. Patients accompanied with other tumors or past medical history of malignancy;
7. Pregnant or lactating patients, all patients participating in this trial must adopt appropriate birth control measures during treatment;
8. Allergic to adriamycin chemotherapy drugs，contrast agent and lipiodol;
9. Patients have poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 3 years
  Overall survival (OS) will be defined as the elapsed time from the enrollment to death from any cause. For surviving patients, follow-up will be censored at the date of last contact (or last date known to be alive). Follow-up for OS will occur every 12 weeks (±1 month) until death or withdrawal of consent from the study.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 3 years
  Progression-free survival (PFS) will be defined as the elapsed time from the first date of study treatment until documented disease progression (as per mRECIST) or death from any cause, whichever is earlier. For patients who remain alive without progression, follow-up time will be censored at the date of last disease assessment.
Adverse event rate | up to 3 years
  Adverse event rate will be defined as the rate of patients who developed adverse event.
Distant metastasis-free survival | up to 3 years
  Progression-free survival (PFS) will be defined as the elapsed time from the first date of study treatment until documented distant metastasis (as per RECIST 1.1) or death from any cause, whichever is earlier. For patients who remain alive without progression, follow-up time will be censored at the date of last disease assessment .

CONTACTS AND LOCATIONS:
Overall Officials: Weijun Fan, M.D, Study Chair — Sun Yat-sen University
Locations (10):
- China (10):
  - Cancer Institute &Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The tumor hospital of Fujian Province, Fuzhou, Fujian
  - the First Affiliated Hospital of SunYat-senUniversity, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Peking University Hospital of Shenzhen, Shenzhen, Guangdong
  - The Second Affiliated Hospital of Shandong University, Jinan, Shandong
  - Shandong Province Hospital, Jinan, Shandong
  - the Affiliated Hospital of Medical College Qingdao University, Qingdao, Shandong
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maida M, Orlando E, Camma C, Cabibbo G. Staging systems of hepatocellular carcinoma: a review of literature. World J Gastroenterol. 2014 Apr 21;20(15):4141-50. doi: 10.3748/wjg.v20.i15.4141. PMID 24764652
- [Background] Bruix J, Sherman M; American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma: an update. Hepatology. 2011 Mar;53(3):1020-2. doi: 10.1002/hep.24199. No abstract available. PMID 21374666
- [Background] Yamashita Y, Taketomi A, Shirabe K, Aishima S, Tsuijita E, Morita K, Kayashima H, Maehara Y. Outcomes of hepatic resection for huge hepatocellular carcinoma (>/= 10 cm in diameter). J Surg Oncol. 2011 Sep 1;104(3):292-8. doi: 10.1002/jso.21931. Epub 2011 Apr 4. PMID 21465490
- [Background] Brunocilla PR, Brunello F, Carucci P, Gaia S, Rolle E, Cantamessa A, Castiglione A, Ciccone G, Rizzetto M. Sorafenib in hepatocellular carcinoma: prospective study on adverse events, quality of life, and related feasibility under daily conditions. Med Oncol. 2013 Mar;30(1):345. doi: 10.1007/s12032-012-0345-2. Epub 2012 Dec 22. PMID 23263829
- [Background] Abdelaziz AO, Nabeel MM, Elbaz TM, Shousha HI, Hassan EM, Mahmoud SH, Rashed NA, Ibrahim MM, Abdelmaksoud AH. Microwave ablation versus transarterial chemoembolization in large hepatocellular carcinoma: prospective analysis. Scand J Gastroenterol. 2015 Apr;50(4):479-84. doi: 10.3109/00365521.2014.1003397. Epub 2015 Jan 16. PMID 25592058
- [Background] Xue T, Le F, Chen R, Xie X, Zhang L, Ge N, Chen Y, Wang Y, Zhang B, Ye S, Ren Z. Transarterial chemoembolization for huge hepatocellular carcinoma with diameter over ten centimeters: a large cohort study. Med Oncol. 2015 Mar;32(3):64. doi: 10.1007/s12032-015-0504-3. Epub 2015 Feb 15. PMID 25682389
- [Background] Min YW, Lee JH, Gwak GY, Paik YH, Lee JH, Rhee PL, Koh KC, Paik SW, Yoo BC, Choi MS. Long-term survival after surgical resection for huge hepatocellular carcinoma: comparison with transarterial chemoembolization after propensity score matching. J Gastroenterol Hepatol. 2014 May;29(5):1043-8. doi: 10.1111/jgh.12504. PMID 24863186
- [Background] Chen MS, Li JQ, Zheng Y, Guo RP, Liang HH, Zhang YQ, Lin XJ, Lau WY. A prospective randomized trial comparing percutaneous local ablative therapy and partial hepatectomy for small hepatocellular carcinoma. Ann Surg. 2006 Mar;243(3):321-8. doi: 10.1097/01.sla.0000201480.65519.b8. PMID 16495695
- [Background] Feng K, Yan J, Li X, Xia F, Ma K, Wang S, Bie P, Dong J. A randomized controlled trial of radiofrequency ablation and surgical resection in the treatment of small hepatocellular carcinoma. J Hepatol. 2012 Oct;57(4):794-802. doi: 10.1016/j.jhep.2012.05.007. Epub 2012 May 23. PMID 22634125
- [Background] Lu MD, Kuang M, Liang LJ, Xie XY, Peng BG, Liu GJ, Li DM, Lai JM, Li SQ. [Surgical resection versus percutaneous thermal ablation for early-stage hepatocellular carcinoma: a randomized clinical trial]. Zhonghua Yi Xue Za Zhi. 2006 Mar 28;86(12):801-5. Chinese. PMID 16681964
- [Background] Huang YH, Wu JC, Chen SC, Chen CH, Chiang JH, Huo TI, Lee PC, Chang FY, Lee SD. Survival benefit of transcatheter arterial chemoembolization in patients with hepatocellular carcinoma larger than 10 cm in diameter. Aliment Pharmacol Ther. 2006 Jan 1;23(1):129-35. doi: 10.1111/j.1365-2036.2006.02704.x. PMID 16393290
- [Background] Kim JH, Won HJ, Shin YM, Kim SH, Yoon HK, Sung KB, Kim PN. Medium-sized (3.1-5.0 cm) hepatocellular carcinoma: transarterial chemoembolization plus radiofrequency ablation versus radiofrequency ablation alone. Ann Surg Oncol. 2011 Jun;18(6):1624-9. doi: 10.1245/s10434-011-1673-8. Epub 2011 Mar 29. PMID 21445671
- [Background] Mizukoshi E, Yamashita T, Arai K, Sunagozaka H, Ueda T, Arihara F, Kagaya T, Yamashita T, Fushimi K, Kaneko S. Enhancement of tumor-associated antigen-specific T cell responses by radiofrequency ablation of hepatocellular carcinoma. Hepatology. 2013 Apr;57(4):1448-57. doi: 10.1002/hep.26153. PMID 23174905
- [Background] Zerbini A, Pilli M, Penna A, Pelosi G, Schianchi C, Molinari A, Schivazappa S, Zibera C, Fagnoni FF, Ferrari C, Missale G. Radiofrequency thermal ablation of hepatocellular carcinoma liver nodules can activate and enhance tumor-specific T-cell responses. Cancer Res. 2006 Jan 15;66(2):1139-46. doi: 10.1158/0008-5472.CAN-05-2244. PMID 16424051
- [Background] Kim YS, Lim HK, Rhim H, Lee MW, Choi D, Lee WJ, Paik SW, Koh KC, Lee JH, Choi MS, Gwak GY, Yoo BC. Ten-year outcomes of percutaneous radiofrequency ablation as first-line therapy of early hepatocellular carcinoma: analysis of prognostic factors. J Hepatol. 2013 Jan;58(1):89-97. doi: 10.1016/j.jhep.2012.09.020. Epub 2012 Sep 27. PMID 23023009
- [Background] Shiina S, Tateishi R, Arano T, Uchino K, Enooku K, Nakagawa H, Asaoka Y, Sato T, Masuzaki R, Kondo Y, Goto T, Yoshida H, Omata M, Koike K. Radiofrequency ablation for hepatocellular carcinoma: 10-year outcome and prognostic factors. Am J Gastroenterol. 2012 Apr;107(4):569-77; quiz 578. doi: 10.1038/ajg.2011.425. Epub 2011 Dec 13. PMID 22158026
- [Background] Peng ZW, Zhang YJ, Chen MS, Xu L, Liang HH, Lin XJ, Guo RP, Zhang YQ, Lau WY. Radiofrequency ablation with or without transcatheter arterial chemoembolization in the treatment of hepatocellular carcinoma: a prospective randomized trial. J Clin Oncol. 2013 Feb 1;31(4):426-32. doi: 10.1200/JCO.2012.42.9936. Epub 2012 Dec 26. PMID 23269991
- [Background] Kim JW, Shin SS, Kim JK, Choi SK, Heo SH, Lim HS, Hur YH, Cho CK, Jeong YY, Kang HK. Radiofrequency ablation combined with transcatheter arterial chemoembolization for the treatment of single hepatocellular carcinoma of 2 to 5 cm in diameter: comparison with surgical resection. Korean J Radiol. 2013 Jul-Aug;14(4):626-35. doi: 10.3348/kjr.2013.14.4.626. Epub 2013 Jul 17. PMID 23901320